CLINICAL TRIAL: NCT07384325
Title: Gravity of Flow: Automating Diuresis
Brief Title: Gravity in Flow: Automating Diuresis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, R.E. Knops, Professor, MD, Amsterdam Universitair Medische Centra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NL84838.018.23; NL-005919 (Registry Identifier: ToetsingOnline (CCMO, Netherlands))
Record Dates: First submitted 2026-01-06; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Automated Urine Monitoring; Urine Output; Fluid Balance; Urinary Catheters; Diuresis
Keywords: Automated urine monitoring; Diuresis monitoring; Indwelling urinary catheter; Fluid balance monitoring

STUDY DESIGN:
Intervention Model Description: Part A: Single-arm technical feasibility using both manual and automated FlowSure monitoring simultaneously. Part B: Two-arm randomized, open-label comparison between manual and automated urine monitoring.
Masking Description: Open-label study; care providers and investigators are aware of group assignment. Data analysis is based on objective device measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Urine Monitoring (Active Comparator): Participants in this arm will be monitored using the standard manual urine measurement system consisting of a measuring chamber and urine collection bag. Nursing staff will manually record hourly urine output in the electronic medical record according to routine hospital procedures.
  Interventions: Device: Manual Urine Monitoring System
- Automated Monitoring (Experimental): Participants in this arm will be monitored using the investigational automated urine output monitoring device. The device continuously weighs the urine collection bag to calculate urine volume in milliliters per hour and automatically transfers data to the electronic medical record.
  Interventions: Device: FlowSure Automated Urine Output Monitor

INTERVENTIONS:
Device: FlowSure Automated Urine Output Monitor — A digital hanging scale that continuously weighs the urine collection bag to determine urine output in milliliters per hour. The device provides real-time diuresis data and automatically transfers measurements to the electronic medical record. FlowSure does not come into contact with the patient or urine and can be reused after surface disinfection.
  Arms: Automated Monitoring
Device: Manual Urine Monitoring System — The current standard-of-care manual urine monitoring system consisting of a measuring chamber and urine collection bag. Nursing staff manually record hourly urine output in the electronic medical record according to routine hospital procedures.
  Arms: Manual Urine Monitoring

SUMMARY:
The goal of this randomized clinical trial is to evaluate the accuracy of automated urine output monitoring using the FlowSure system compared to standard manual urine monitoring in hospitalized patients with an indwelling urinary catheter.

The main questions it aims to answer are:

How accurate is the automated FlowSure monitoring compared with manual urine monitoring over defined time intervals (8-hour nursing shifts and 24-hour periods)?

Does the automated system improve completeness of hourly urine output registration compared with manual documentation?

Researchers will compare patients monitored with the automated FlowSure device to those monitored using the manual method to determine whether automation provides more accurate and complete diuresis data.

Participants will:

Be adult patients admitted to the hospital with a urinary catheter inserted for routine medical reasons (not related to this study).

In Part B, be randomized to either manual urine monitoring or automated FlowSure monitoring for defined time intervals.

There is no direct benefit to participants. The potential societal benefit lies in improving the accuracy, efficiency, and safety of diuresis monitoring through automation. The risks are minimal and limited to use of the FlowSure device in addition to, or instead of, standard monitoring; no additional procedures are performed.

DETAILED DESCRIPTION:
Accurate monitoring of urine output is essential in the management of hospitalized patients, particularly those with hemodynamic instability or fluid balance disorders. Currently, diuresis monitoring is performed manually by nursing staff, which is labor intensive and prone to transcription or timing errors. The FlowSure system is an automated urine output monitoring device designed to continuously measure and record urine production and transfer these data directly to the electronic medical record (EMR). Automation may improve data quality, reduce nursing workload, and enhance patient safety.

This study consists of two parts. Part A is a technical feasibility study in which patients are simultaneously monitored using both manual and automated FlowSure systems to evaluate concordance between the two methods under real-world conditions. Part B is a two-arm randomized, non-blinded intervention study comparing automated versus manual urine output monitoring. Patients will be randomized in a 1:1 ratio to either standard manual monitoring or automated FlowSure monitoring. Randomization occurs after insertion of a urinary catheter, which is placed for medical reasons unrelated to the study.

The primary objective of Part B is to assess the accuracy of urine production measurement by the automated FlowSure monitor compared with manual monitoring over two time frames: (1) an 8-hour nursing shift and (2) a full 24-hour period. The primary endpoint is the completeness and accuracy of hourly diuresis registration between the two monitoring methods. Secondary analyses will include evaluation of data recording efficiency and the rate of missing or incorrect entries in the EMR.

There is no direct therapeutic benefit to participants. The anticipated scientific and societal benefit lies in improving the reliability and efficiency of diuresis monitoring, potentially enhancing patient care and reducing nursing workload. The risks associated with participation are minimal. In Part A, the automated monitor operates in addition to the manual system; in Part B, patients are monitored using only one method. In case of device malfunction or data loss, urine output can be estimated from total collected volume over time. Given the low risk profile and the potential to improve clinical monitoring practices, the overall risk-benefit balance of the study is considered favorable.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Currently hospitalized.
* Indwelling urinary catheter inserted for medical reasons unrelated to the study.
* Able and willing to provide written informed consent.
* No specific urological problems.

Exclusion Criteria:

* No urinary catheter in place.
* Diuresis < 30 mL per hour at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Accuracy of urine output measurement using the FlowSure automated monitoring device compared with manual monitoring | Over a single 8-hour nursing shift and a full 24-hour monitoring period
  Accuracy will be defined as the agreement between urine output measured by the FlowSure device and manual measurement (reference standard) over predefined time intervals of 8 hours and 24 hours.

SECONDARY OUTCOMES:
Completeness of hourly urine output registration in the electronic medical record | Over a single 8-hour nursing shift and a full 24-hour monitoring period
  Percentage of expected hourly urine output entries successfully recorded in the electronic medical record during the 8-hour and 24-hour measurement periods.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Brouwer, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Locatie AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data because this is a single-center device validation study with limited sample size. Aggregated results will be published in peer-reviewed journals.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT07384325/Prot_SAP_000.pdf